CLINICAL TRIAL: NCT03948009
Title: TREatment of Uretral STRICTure With Self-catheterization : Tolerance Evaluation
Acronym: TRESTRICTT
Status: Terminated | Type: Observational
Why Stopped: The investigator did not have enough time to manage the study.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7292
Record Dates: First submitted 2018-11-22; First posted 2019-05-13 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2020-08

CONDITIONS: First or Second Uretral Stenosis; Diagnosed With Uretral Fibroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urethral stenosis has a recurrent character. The clean intermittent self-catheterization can be proposed for repeat stenosis. This study seeks to explore the tolerance of clean intermittent self-catheterization in the evolution of urethral stenosis after urethrotomy.

ELIGIBILITY:
Inclusion criteria:

* Men between 18 and 80
* First or second uretral stenosis, diagnosed with uretral fibroscopy

Exclusion criteria:

* Not multiple, strength or long stenosis
* No previous surgery of the urethra
* Refusal to participate to the study
* Inability to perform self-catheterization

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men between 18 and 80 First or second uretral stenosis, diagnosed with uretral fibroscopy
  Not multiple, strength or long stenosis No previous surgery of the urethra
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Number of patient which continue clean intermittent self-catheterization. | 18 months
  Evaluation of patients tolerance with clean intermittent self-catheterization

SECONDARY OUTCOMES:
Comparaison of uroflowmetry | 18 months
  Evaluation of patients urinary profile
Comparaison of Urinary Score Profile (USP) | 18 months
  Evaluation of patients quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Thibault TRICARD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided